CLINICAL TRIAL: NCT00911079
Title: Pilot Study of a Catheter-based Ultrasound Hyperthermia System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, I-Chow Hsu, Professor, Radiation Oncology, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CDR0000643085; 08992 (Other: University of California, San Francisco); 5R01CA122276 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Cervical Cancer; Prostate Cancer
Keywords: Stage III, IV cervical cancer; Rising prostate specific antigen (PSA) after local therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hyperthermia with HDR brachytherapy (Experimental): Hyperthermia will be delivered within approximately 2 hours of (HDR) brachytherapy associated with the implant session
  Interventions: Procedure: Hyperthermia; Radiation: HDR brachytherapy

INTERVENTIONS:
Procedure: Hyperthermia — Single course of Catheter-based Ultrasound Hyperthermia (within approximately 2 hours of a Standard-of-care High Dose Rate (HDR) Brachytherapy)
Radiation: HDR brachytherapy — Completion of standard-of-care high dose rate (HDR) Brachytherapy treatments (radiation fractions) using Session #1 catheter implants

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Ultrasound energy may be able to kill tumor cells by heating up the tumor cells without affecting the surrounding tissue. Implant radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving ultrasound hyperthermia therapy after implant radiation therapy may kill more tumor cells.

PURPOSE: This clinical trial is studying ultrasound hyperthermia therapy to see how well it works after implant radiation therapy in treating patients with Stage III/IV cancer of the cervix or prostate cancer with a rising prostate specific antigen (PSA) after prior local therapy.

DETAILED DESCRIPTION:
OUTLINE: Patients undergo standard high-dose rate (HDR) brachytherapy. Approximately 2 hours after brachytherapy, patients undergo catheter-based ultrasound hyperthermia therapy over 60 minutes. Treatment with HDR brachytherapy and hyperthermia therapy repeats within 1-3 weeks. Patients may then undergo 2 additional standard HDR brachytherapy sessions.

After completion of study therapy, patients are followed at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to be given HDR brachytherapy for treatment of solid tumor of the following:

  * Cervical cancer Stage III or IV OR
  * Prostate cancer (with rising prostate specific antigen after prior local therapy)
* Age >=18 years
* Eligible for brachytherapy as determined per clinical standard of care.
* Ability to give written informed consent and willingness to comply with the requirements of the protocol

Exclusion Criteria:

* Patients who are not candidates for HDR brachytherapy
* Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-12-18 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-related toxicities by treatment type | Up to 3 months
  All patients treated with at least one hyperthermia session will be included in the safety analysis. The frequency by grade for all treatment-related adverse events will be tabulated by type as classified in NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 and presented separately for the first and second hyperthermia treatments.
Frequency of treatment-related toxicities by accrual plan | Up to 3 months
  All patients treated with at least one hyperthermia session will be included in the safety analysis. The frequency by grade for all treatment-related adverse events will be tabulated by type as classified in NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 presented for the 2 subsets of patients corresponding to the plan for accrual: the first 3 patients with gynecologic cancer, then the final 9 patients with gynecologic cancer; and the first 3 patients with prostate cancer, then the final 9 patients with prostate cancer
Proportion of patients treated according to the specified temperature and timing criteria. | Up to 4 weeks
  The feasibility of administering hyperthermia to patients receiving standard brachytherapy will be summarized by the proportion of patients completing the treatment as planned. The proportion and 95% confidence interval will be calculated for each of the two hyperthermia sessions

SECONDARY OUTCOMES:
Average maximum prostate temperature (Tmax) | Up to 4 weeks
  Attainable temperature and thermal dose distributions will be summarized using descriptive statistics and presented separately for each hyperthermia treatment
Minimum temperature (Tmin) | Up to 4 weeks
  Attainable temperature and thermal dose distributions will be summarized using descriptive statistics and presented separately for each hyperthermia treatment
Median temperature (T50) | Up to 4 weeks
  Attainable temperature and thermal dose distributions will be summarized using descriptive statistics and presented separately for each hyperthermia treatment
Number of times temperature exceeded by 90% of the measured temperature points (T90) | Up to 4 weeks
  Attainable temperature and thermal dose distributions will be summarized using descriptive statistics and presented separately for each hyperthermia treatment
Cumulative Equivalent Minutes at 43 degree celsius (ºC) for 90% of the measured points (CEM43T90) | Up to 4 weeks
  Attainable temperature and thermal dose distributions will be summarized using descriptive statistics and presented separately for each hyperthermia treatment

CONTACTS AND LOCATIONS:
Overall Officials: I-Chow J. Hsu, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT00911079/ICF_000.pdf